CLINICAL TRIAL: NCT03734003
Title: Evaluation of Controllable Infrared Bioeffect Effect for the Treatment of Cutaneous Warts After 3 Months: a Multicenter, Randomized, Open Label Controlled Trial
Brief Title: Infrared Bioeffect System for the Treatment of Cutaneous Warts
Acronym: wart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH20180726
Record Dates: First submitted 2018-07-30; First posted 2018-11-07 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2019-06

CONDITIONS: Cutaneous Warts; Human Papilloma Virus
Keywords: hyperthermia; human papilloma virus; cutaneous warts
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controllable infrared bioeffect system for cutaneous warts (Experimental): Controllable infrared bioeffect system at 44±2℃ for 30 mins on target lesion, at days of 1, 2, 3, 15, 16, 23, 30.
  Common warts, plantar warts, and condyloma acuminata
  Interventions: Device: controllable infrared bioeffect system
- Liquid nitrogen cryotherapy for cutaneous warts (Active Comparator): Liquid nitrogen crytotherapy at days 1, 15, 30.
  Interventions: Device: liquid nitrogen

INTERVENTIONS:
Device: liquid nitrogen — As an active comparator, for patients with cutaneous warts, liquid nitrogen crytherapy is applied
  Arms: Liquid nitrogen cryotherapy for cutaneous warts
Device: controllable infrared bioeffect system — As an experimental arm, for patients with cutaneous warts
  Arms: Controllable infrared bioeffect system for cutaneous warts

SUMMARY:
Local hyperthermia at 44℃ can promote some alterations of immulogical indicators. The procedure is convenient in clinic, has high tolerance with less trauma and less pain. Based on domestic and abroad clinical practice, the investigators observed initially that local hyperthermia brought great benefits to cutaneous warts. In comparison with liquid nitrogen, the safety and efficacy of controllable infrared bioeffect system to treat skin disease has been evaluated. This proved it could be used in treatment of skin warts, and clinical trial met the requirements of Standards for quality control of clinical trials on medical devices, and can be used in product registration and declaration.

DETAILED DESCRIPTION:
Mild local Hyperthermia with a certain temperature range has been successfully used in the treatment of some diseases. It has been utilised in the treatment of some neoplasm, fungal and HPV infections. Investigators' study found that local hyperthermia at 44°C could cleared HPV in more than half of the patients with plantar warts. Investigators also note the fact that in patients with multiple lesions, the clearance of the target lesion is commonly followed by clearance of other distant lesions, a phenomenon suggesting that local hyperthermia could aid in establishing a specific immune response to eliminate HPV.So the purpose of the study is to evaluate the safety and efficacy of controllable infrared bioeffect system to treat cutaneous warts. This trial was designed into two groups, one was experimental group (thermal therapy group), the other one was control group (liquid nitrogen cryotherapy group). The ratio of participants was 1:1 in experiment group and control group. The main evaluation indicator was the recovery rate after 4 months of initial treatment.

ELIGIBILITY:
Inclusion Criteria :

18-70 years old signed informed consent clinical diagnosed HPV induced cutaneous warts no local or systemic therapy within 3 months effective contraception for 6 months after signed informed consent

Exclusion Criteria:

HbsAg(+), HCV-Ab(+), HIV-Ab(+) skin lesions associated with other infections pregnant or breast-feeding woman unsuitable to be treated by liquid nitrogen cryotherapy scar diathesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Recovery rate of cutaneous warts | 3 months after the last time of treatment
  to evaluate the clearance rate in different treatment groups 3 months after treatment

SECONDARY OUTCOMES:
Clearance rate of target lession | 3 months after the last time of treatment
  to evaluate the recovery rate of target lession in different treatment groups 3 months after treatment
Clearance rate of non-target lession | 3 months after the last time of treatment
  to evaluate the recovery rate of non-target lession in different treatment groups 3 months after treatment
the visual analogue score (VAS) of pain | 3 months after the last time of treatment
  to evaluate the score of VAS (0 score represents no pain; 10 score represents sharp pain) in different treatment groups 3 months after treatment
Clearance rate of virus | 3 months after thelast time of treatment
  to evaluate the clearance rate of virus in different treatment groups 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Study Director — No. 1 Hospital of China Medical University
Locations (1):
- No. 1 Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi RQ, Zhou J, Xiao B, Xu H, Qiao S, Zhu P, Xia L, Yang Y, Zhang L, Yan H, He C, Sun Y, Niu X, Zhang Y, Fu L, Wang X, Chen HD, Li S, Gao XH. Reprint of: Clearance of multiple cutaneous warts by targeting a single lesion: A randomized comparative evaluation of mild local hyperthermia versus cryotherapy. J Am Acad Dermatol. 2023 Mar;88(3):647-649. doi: 10.1016/j.jaad.2023.02.001. Epub 2023 Feb 18. No abstract available. PMID 36804149